CLINICAL TRIAL: NCT03483597
Title: The Survey of Satisfaction in Chinese Rheumatologists and Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Chinese SLE Treatment And Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: CRDC-satisfaction
Record Dates: First submitted 2018-03-21; First posted 2018-03-30 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2018-03

CONDITIONS: Rheumatoid Arthritis; Satisfaction
MeSH Terms: conditions — Arthritis, Rheumatoid; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- rheumatologists: Inclusion criteria: Registered rheumatoid specialist physicians subordinated to the 12 designated hospitals The Treatment Satisfaction Questionnaire for Medication (TSQM-II) will be used in rheumatologists.
  Interventions: Other: TSQM-II
- patients: Inclusion criteria: Aged over 18, confirming RA for more than 6 months Exclusion criteria. Patients with Chinese reading comprehension barriers (unable to complete the questionnaire independently), without any RA treatment The Treatment Satisfaction Questionnaire for Medication (TSQM-II) will be used in patients.
  Interventions: Other: TSQM-II

INTERVENTIONS:
Other: TSQM-II — Treatment Satisfaction Questionnaire for Medication (TSQM Version II) will be used in all groups

SUMMARY:
A questionnaire for this research is designed, which initiated from TSQM-II treatment satisfaction questionnaire and based on research launched by rheumatology and immunology departments of Chinese 12 public tertiary hospitals distributed directionally by Chinese Rheumatism Data Center (CRDC). The research is about treatment satisfaction and its influencing factors for Chinese rheumatoid immunologists and rheumatoid arthritis (RA) patients as well as their expectations for treating this disease. This research will explore the matching degree between treatment satisfaction and expectation about rheumatoid arthritis from doctors and patients.

DETAILED DESCRIPTION:
In the last decade, China has made quick progress on treatment of rheumatoid arthritis. However, the improvement of remission rate cannot fully represent needs of patients for health. To meet health demands of patients and improve their satisfaction, an efficacy evaluation system based on the outcome report of patients should be established. A questionnaire for this research is designed and mended in view of TSQM-II treatment satisfaction questionnaire and the actual situation of RA diagnosis and treatment in China. An investigation on treatment satisfaction and its influencing factors for Chinese rheumatoid immunologists and rheumatoid arthritis (RA) patients as well as their expectations for this disease is carried out based on 120 rheumatoid immunologists and 1,200 rheumatoid arthritis patients (1:10) from Chinese 12 public tertiary hospitals distributed directionally by Chinese Rheumatism Data Center (CRDC). The research concludes rheumatoid specialist physicians for doctor population, and persons aged over 18 for patient population who has been confirmed as RA for 6 months above, excluding patients with Chinese reading comprehension barriers or without any RA treatment. Finally, summarize and analyze the total score of satisfaction from doctors and patients, average score of doctors and patients for various medical demands, as well as the satisfaction of patients about communication and service during medical treatment.

ELIGIBILITY:
Inclusion Criteria:

Doctors - registered rheumatoid specialist physicians subordinated to the 12 designated hospitals Patients - aged over 18, confirming RA for more than 6 months

Exclusion Criteria:

Doctors - N/A Patients - with Chinese reading comprehension barriers (unable to complete the questionnaire independently), without any RA treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects come from 12 hospitals in Chinese Rheumatism Data Center.
Sampling Method: Non-Probability Sample
Enrollment: 1365 (Actual)
Dates: Start 2018-03-31 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Total score of patient satisfaction | 1 day
  Total score of patient satisfaction

SECONDARY OUTCOMES:
Average score of patients for various treatment demands | 1 day
  Average score of patients for various treatment demands
Average score of patients for long-term treatment demands | 1 day
  Average score of patients for long-term treatment demands
Average score of patients for new drug demands | 1 day
  Average score of patients for new drug demands
Total score of doctor satisfaction | 1 day
  Total score of doctor satisfaction
Average score of doctors for various treatment demands | 1 day
  Average score of doctors for various treatment demands
Average score of doctors for long-term treatment demands | 1 day
  Average score of doctors for long-term treatment demands
Average score of doctors for new drug demands | 1 day
  Average score of doctors for new drug demands

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, Doctor, Study Chair — Director of Rheumatology and Immunology Department Chinese Academy of Medical Sciences &Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No